CLINICAL TRIAL: NCT04853290
Title: Patient Experience With Ultrasound-guided Versus Conventional Peripheral Venipuncture: a Randomized Clinical Trial
Brief Title: Patient Experience in Peripheral Venipuncture With and Without Ultrasound
Acronym: PERCEPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 40240920.6.0000.5327
Record Dates: First submitted 2021-04-16; First posted 2021-04-21 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Peripheral Venous Catheterization; Ultrasonography; Pain
Keywords: Peripheral venous catheterization; Ultrasonography; Pain; Patient satisfaction; Nursing; Clinical trial
MeSH Terms: conditions — Pain; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: It is a PROBE (Prospective Randomized Open Blinded End Point), parallel, controlled, and single center randomized clinical trial (RCT).
Who Masked: Investigator, Outcomes Assessor
Masking Description: Researchers and investigators responsible for data collection will be blinded for collection and analysis of data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Ultrasound-guided peripheral venipuncture performed by a registered nurse with expertise in vascular access.
  Interventions: Device: Ultrasound-guided peripheral venipuncture
- Control group (Active Comparator): Conventional peripheral venipuncture performed by a registered nurse from a clinical inpatient unit.
  Interventions: Device: Conventional peripheral venipuncture

INTERVENTIONS:
Device: Ultrasound-guided peripheral venipuncture — Ultrasound-guided peripheral venipuncture performed by a proficient vascular access registered nurse. The procedure will be performed according to the standard operational protocol for ultrasound guided peripheral venipuncture instituted at the hospital where the study will be conducted. Site Rite 8 or Site Rite 5 ultrasound machines (Bard Access Systems, Inc., USA) will be used on the procedures.
  Arms: Intervention group
Device: Conventional peripheral venipuncture — Conventional peripheral venipuncture performed by the registered nurse at the clinical inpatient unit. The procedure will be performed according to the standard operational protocol for peripheral venipuncture protocol instituted in the hospital where the study will be conducted
  Arms: Control group

SUMMARY:
Randomized clinical trial to compare the patient's experience after peripheral venipuncture catheterization using the conventional technique (vein visualization and palpation) versus ultrasound-guided venous puncture.

Patients with indication of peripheral venous puncture, admitted to the clinical inpatient units on the hospital where the study will be conducted (Hospital de Clinicas de Porto Alegre - HCPA) will be enrolled in this single-center trial and will be randomized to conventional peripheral venipuncture performed by a registered nurse; or ultrasound-guided peripheral venipuncture performed by a registered nurse with expertise in vascular access.

DETAILED DESCRIPTION:
Study Protocol

When there is a need of a peripheral venous access for the inpatient, the medical or nursing care team will contact the researchers, informing the personal data of the possible candidate to participate in the study. By fulfilling the eligibility criteria, the patient will be invited and informed about the study proposal; and, if he agrees to participate, he will sign the consent form. The type of procedure to be performed will be randomized through a draw. The procedure options are:

1. Intervention: ultrasound peripheral venipuncture executed by specialized nurses (vascular access program), or
2. Control: conventional peripheral venipuncture executed by clinical practice nurses..

Individuals who do not agree to participate in the study will have their data stored on a patient exclusion checklist. In both groups, intervention and control, up to two attempts will be made by the same professional and, if there is no success on the procedure, another professional will be designated for two more attempts. Ultrasound Site Rite 8 or Ultrasound Site Rite 5, which are portable ultrasound devices that include 2D ultrasound imaging in real time, will be used on the Intervention Group (1) procedure.

The peripheral venipuncture procedure for both groups will be performed according to the standard operating procedures recommended by the institution where the study will be conducted (HCPA). The catheters to be used will be the peripheral venous catheters made available by the institution.

If there is a failure of puncture in the Control Group (2), the study participant will follow the institution's routine to adapt an appropriate vascular access, which is the activation of a nurse specialist in vascular access, who can perform peripheral venipuncture guided by ultrasound. In the event of a new insertion failure, the care team (doctor and nurse) discusses the case to define a new approach according to the infusional therapy, considering the protocol for the indication of venous vascular accesses at the institution. Thereafter, the patient can proceed for oral treatment, insertion of a peripherally inserted central catheter, insertion of a short-term central venous catheter, hypodermoclysis, long-term central venous catheter (totally or semi-implanted), according to the decision of the assistant team.

In the case of failure of the puncture in the Intervention Group (1), the study participant will follow the same routine of the institution, as explained above, for the adequacy of an adequate vascular access. However, in this case, the nurse specialist in vascular access will not be contacted, as the intervention procedure already uses ultrasound.

All participants who successfully insert a peripheral venous catheter in both groups will be monitored for the occurrence of any event related to the procedure from the time of insertion of the catheter until the loss of access for any reason, removal of the device at the end of therapy, discharge, death or eight days of follow-up, whichever comes first. Peripheral venous access that remains for more than eight days will be counted as event-free, access survival. Study participants with failed insertion will have the outcome computed in the database and will be followed up for another 48 hours to assess any complications resulting from the puncture attempt.

ELIGIBILITY:
Inclusion Criteria:

* Adults, age = or > 18 years;
* Admitted to the clinical inpatient units on the hospital where the study will be conducted (HCPA), with indication of peripheral venous puncture;
* Patients who do not configure emergency care.

Exclusion Criteria:

* Patients who have already received ultrasound-guided peripheral venipuncture at the current hospitalization;
* Patients in a critical or unstable clinical condition;
* Patients admitted to surgical units at HCPA;
* Patients in coronavirus (COVID-19) care units.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2021-09-23 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Patient's experience of pain during the procedure | up to 5 minutes.
  Patient's experience of pain during the procedure of peripheral venipuncture, evaluated immediately after the procedure using the 10 cm verbal Numerical Rating Scale (vNRS). The response indicated by the patient regarding the degree of felt pain during the procedure, from 0 to 10, with 10 being the most intense pain, will be computed.
Patient's experience with the method used to obtain venous access (1/2) | up to 5 minutes.
  Patient's experience with the method used to obtain venous access, assessed using the Net Promoter Score (NPS), a single metric instrument that quantifies the answers to a single direct research question: "How likely are you to recommend this procedure?". Three categories of respondents are identified and classified as 'promoters' (those who would definitely recommend), 'passive' (who are widely satisfied, but would not recommend) and 'detractors' (who actively discourage others from trying the procedure).
Patient's experience with the method used to obtain venous access (2/2) | up to 10 minutes.
  Additionally, it will be assessed the elements: a) patient emotional aspect during the procedure (anxiety, discomfort, importance of the procedure, fear, concern, safety); b) venous catheter insertion site; c) number of venipuncture attempts; d) dressing and device fixation on the skin; e) procedure's time duration; as relevant indicators for the characterization of the procedure as a positive or a negative experience for the patients. Data will be computed using a 10 point Likert scale score, in which 1 point rates the worst experience and 10 points an excellent experience.

SECONDARY OUTCOMES:
Peripheral intravenous catheter dwell time | Daily monitoring, until catheter removal
  Accesses that remained functional, intact, fixed and without phlogistic signs when the device was inserted into the skin were considered durable.
Complications during the vascular access device permanence | Daily monitoring, up 2 days after catheter removal
  Complications that might occur during the permanence of the vascular access device (phlebitis, obstruction, leakage, infiltration, etc), measured through clinical assessment. In the case of the development of phlebitis, it will be evaluated through the application of the Visual Infusion Phlebitis Scale (from the Infusion Nurses Society), which classifies the lesion up to five degrees, according to the progression and severity of the signs and symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Eneida R Rabelo-Silva, RN, MSc, ScD, Principal Investigator — Hospital de Clinicas de Porto Alegre
Locations (1):
- Universidade Federal do Rio Grande do Sul - Post Graduated Program, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tada M, Yamada N, Matsumoto T, Takeda C, Furukawa TA, Watanabe N. Ultrasound guidance versus landmark method for peripheral venous cannulation in adults. Cochrane Database Syst Rev. 2022 Dec 12;12(12):CD013434. doi: 10.1002/14651858.CD013434.pub2. PMID 36507736